CLINICAL TRIAL: NCT00463216
Title: A Coordinated Return to Work Program for Workers on Long-term Sickness Absence Due to Musculoskeletal Disorders: a Prospective Controlled Intervention Study
Brief Title: A Coordinated Return to Work Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: F03-05
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2007-03

CONDITIONS: Back Pain
Keywords: back, neck, pain, sick leave
MeSH Terms: conditions — Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: A multidisciplinary diagnostic evaluation

SUMMARY:
The aim of the study is to investigate the possibility that a diagnostic evaluation by a multidisciplinary team reduces the length of sick leave.

DETAILED DESCRIPTION:
Workers on sick leave due to back, neck or shoulder pain are randomized into 2 groups. Individuals in the intervention group are offered an extra multidisciplinary diagnostic evaluation. The multidisciplinary team consists of an occupational physician, a physiotherapist, a chiropractor, a psychologist and a social worker. The result is a coordinated evaluation of the individuals problems with suggestions as to further actions. The focus is on evaluating, if and when the individual can return to work. No treatment is given.

Verbatim exemption from the local medical ethics board:

"February 19, 2004 Journal no. VF 20040030 JK/csf Re: research project: A Coordinated Return to Work Program (KIA) The The Medical Ethics Committee of Vejle and Funen Counties has reviewed this research project at its meeting on February 9, 2004.

The entire committee decided that this project is an HTA (Health Technology Assessment) study and not a biomedical research project.

Therefore the committee decided that the project is not within the committee's legal competence areas, and is exempt from approval by a medical ethics committee before being carried out.

The committee has no further comments to this case. on behalf of the committee Sincerely Erik Laier Jette Krarup

__________________________________________________________________________________________________________________________________________________

Odense University Hospital direct telephone: +45 6541 3425 Kløvervaenget 10, 2.sal e-mail: Vejle-fynkomiteen@ouh.fyns-amt.dk 5000 Odense C fax: +45 6619 4392 Denmark"

ELIGIBILITY:
Inclusion Criteria:

* On sick leave due to back,
* Shoulder or neck pain

Exclusion Criteria:

* Pregnant,
* Other causes of sick leave

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-04; Study Completion 2006-04

PRIMARY OUTCOMES:
Number of hours on sick leave in the 1 year study period

SECONDARY OUTCOMES:
Sick leave related costs

CONTACTS AND LOCATIONS:
Overall Officials: Jorgen Kilsgaard, chiropract, Principal Investigator — Vejle County, Vejle, Denmark
Locations (1):
- Dept Occup Environ Med, Vejle Hospital, Vejle, Vejle, Denmark